CLINICAL TRIAL: NCT05334654
Title: Bivalirudin Versus Enoxaparin for Anticoagulation in Critically Ill COVID-19 Patients: a Pilot Randomized Controlled Trial
Brief Title: Bivalirudin Versus Enoxaparin in Critically Ill COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Director of the Intensive Care and Anesthesia Department, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Bivalirudin COVID-19
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Acute Respiratory Failure; SARS CoV 2 Infection; Anticoagulants
MeSH Terms: conditions — COVID-19 | interventions — enoxaparin sodium; bivalirudin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators and Outcome assessors will not take part in the care of patients. Data will be provide in anonymous form without any indication to the assigned treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enoxaparin sodium (Active Comparator): Enoxaparin sodium twice daily, according to the renal function and clinical indication
  Interventions: Drug: Enoxaparin Sodium
- Bivalirudin (Experimental): Bivalirudin will be administered by continuous infusion, until day 7. Bivalirudin will be administered at dosage of 0,25 mg/kg in first 30 minutes, followed by continuous infusion of 0,2 mg/kg/h until 7 days. The infusion rate will be adjusted targeting a prothrombin time ratio of about 1.5.
  Interventions: Drug: Bivalirudin

INTERVENTIONS:
Drug: Enoxaparin Sodium — Enoxaparin will be subcutaneously administered at a dosage from 4000 to 8000 twice daily according
  Arms: Enoxaparin sodium
Drug: Bivalirudin — Bivalirudin will be intravenously administered to obtain an activated prothrombin time (aPTT) of 1.5 fold of the normal values.
  Arms: Bivalirudin

SUMMARY:
Coronavirus Disease (COVID-19) is characterized by a hypercoagulable state, sometimes difficult to be managed with heparin. Bivalirudin, a member of the direct thrombin inhibitor drug class, offers potential advantages compared to heparin, including to its ability to exert its effect by directly attaching to and inhibiting freely circulating and fibrin-bound thrombin.

Investigators have therefore designed this pilot open-label randomized controlled trial to assess if a off-label infusion of bivalirudin may reduce thrombosis, mortality, Intensive Care Unit (ICU) length of stay and increase ventilator free days of patients admitted in ICU for acute respiratory failure due to COVID-19, as compared to first-line treatment with heparin.

ELIGIBILITY:
Inclusion Criteria:

* ratio between arterial partial pressure to inspired fraction of oxygen (PaO2/FiO2) < 200 mmHg
* age equal or greater of 18 years/old
* detection of coronavirus 2019 at the nasal swab;
* need for endotracheal intubation and invasive mechanical ventilation

Exclusion Criteria:

* known allergies to one of the two investigated drugs
* presence of hematological diseases
* pregnancy
* recent (10 days) surgery
* presence of active bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Time spent under invasive mechanical ventilation | from randomization till 28 days after randomization
  number of days that patient would require invasive mechanical ventilation

SECONDARY OUTCOMES:
Incidence of vein thrombosis and embolism | from randomization till 28 days after randomization or ICU discharge
  Number of patients with diagnosis of deep vein thrombosis and/or pulmonary embolism
Gas Exchange | Every day till 28 days after randomization or ICU discharge
  Daily evaluation of oxygenation through arterial blood gases
Intensive Care Unit length of stay | Up to 1 year
  Number of days spent in Intensive Care Unit
Intensive Care Unit mortality | Up to 1 year
  Number of patients died during the Intensive Care Unit stay

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Magna Graecia University
Locations (1):
- AOU Mater Domini, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
The individual patients data will be shared only after the publication of the study on an international peer-reviewed journal and on scientific and intelligible proposal
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after publication on an indexed international and peer-reviewed journal
Access Criteria: Access will be allowed after contacting by email the principal investigator, by providing and intelligible and scientific proposal